CLINICAL TRIAL: NCT01644864
Title: Can Post-operative TAP Block Improve Quality of Recovery After C-sections in Patients on Methadone Maintenance Therapy for Opioid Abstinence?
Brief Title: Can Post-operative TAP Block Improve Quality of Recovery After C-sections in Patients on Methadone Maintenance?
Acronym: TAP
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No participants were enrolled. The PI left the institution.
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 12D.37
Record Dates: First submitted 2012-07-17; First posted 2012-07-19 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Uncontrolled Postoperative Pain
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): saline injection
  Interventions: Drug: placebo
- Experimental (Experimental): 0.375% ROPIVACAINE
  Interventions: Drug: 0.375% ROPIVACAINE

INTERVENTIONS:
Drug: 0.375% ROPIVACAINE
  Arms: Experimental
Drug: placebo
  Arms: Placebo

SUMMARY:
This is a prospective randomized double-blind placebo controlled study (0.375% Ropivacaine vs. 0.9% saline) designed to evaluate the effectiveness of transverse abdominis plane (TAP) block in the first 48 hours after c-section in patients receiving methadone therapy. The TAP block will be performed by a regional anesthesiologist in the operating room after delivery of the baby.

DETAILED DESCRIPTION:
Introduction:

Cesarean sections are the most common surgical operations performed in the U.S (1). Patients requiring c-section who are on methadone maintenance often have uncontrolled pain due to opioid tolerance. The current treatment is to utilize large amounts of opioids via PCA thus resulting in a challenging situation with poor patient satisfaction.

The Transversus abdominis plane (TAP) block has been studied with success in many abdominal surgeries including c-sections (2-5). The anterior abdominal wall is innervated by anterior divisions of spinal segmental nerves which lie between the transversus abdominis and internal oblique muscle layers. Blockade of these nerves with local anesthetics may last up to 24 hours. There have been no efficacy studies performed using the TAP block in patients receiving chronic methadone maintenance undergoing c-sections.

Methods:

This is a prospective randomized double-blind placebo controlled study (0.375% Ropivacaine vs. 0.9% saline) designed to evaluate the effectiveness of transverse abdominis plane (TAP) block in the first 48 hours after c-section in patients receiving methadone therapy. The TAP block will be performed by a regional anesthesiologist in the operating room after delivery of the baby.

Objective:

The primary objective of this study is to measure pain levels after c-sections in patients receiving methadone therapy utilizing visual analog scale (VAS) and assessing opioid consumption during the first 48 hours compared to placebo.

Conclusion:

It is hypothesized that patients receiving TAP block will have decreased pain intensity and less opioid consumption during the first two postoperative days compared to placebo. Therefore we believe postoperative TAP block to be an effective adjuvant to pain control for patients on methadone maintenance following c-section.

ELIGIBILITY:
Inclusion Criteria:

* Laboring patients will only be enrolled in the study if they have a c-section performed. Inclusion criteria include patients who are 18-40 yr of age, ASA physical status I-III, 50-100 kg, 150 cm tall or greater, and English-speaking

Exclusion Criteria:

* Patient refusal, methadone use for chronic pain, contraindications to administration of regional anesthesia (e.g., allergy to a local anesthetic, local infection and coagulopathy), significant neurologic disorders of the lower extremity, and psychiatric or cognitive disorders.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-07; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Quality of Recovery after TAP block | 48 hours
  The primary objective of this study is to measure pain levels after c-sections in patients on methadone maintenance therapy for opioid abstinence. Our objectives are to evaluate the onset and extent of the sensory block following TAP block with 40 mL 0.375% ropivacaine injection compared to placebo block. The degree of sensory block will determine quality of pain scores and degree of opioid consumption. The secondary objective is to administer a previously validated quality of recovery scale (QoR-40) on post-operative days 1 & 2 (POD 1 & 2).

CONTACTS AND LOCATIONS:
Overall Officials: Kishor Gandhi, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States